CLINICAL TRIAL: NCT05827458
Title: An Adequate Cost Effective Follow Up Protocol For Bone and Soft Tissue Sarcomas: - A Prospective Randomized Trial
Brief Title: An Adequate Cost Effective Follow Up Protocol For Bone and Soft Tissue Sarcomas
Acronym: TOSS
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Terry Fox Foundation (Other)
Responsible Party: Principal Investigator, Ajay Puri, Professor, Tata Memorial Hospital
Other Study IDs: TMH BST-216
Record Dates: First submitted 2013-02-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Sarcomas
Keywords: bone tumor; soft tissue tumor; cancer
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Soft Tissue Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- I A: INTENSIVE 3 MONTHS Appropriate local imaging including ultrasound for soft-tissue sarcomas at three-month follow-up A CT scan of the chest was done on a six-monthly basis. CXR at the intervening three-month follow-up.
- I B: INTENSIVE 6 MONTHS
  Appropriate local imaging including ultrasound for soft-tissue sarcomas at six month follow-up A CT scan of the chest was done on a six-monthly basis
- II A: COST EFFECTIVE 3 MONTHS Appropriate local imaging including ultrasound for soft-tissue sarcomas at three-month follow-up with CXR
- II B: COST EFFECTIVE 6 MONTHS Appropriate local imaging including ultrasound for soft-tissue sarcomas at six month follow-up with CXR

SUMMARY:
Bone and soft tissue sarcomas are rare tumors, accounting for approximately 1% of all adult malignancies. The majority of bone and soft tissue sarcomas occur in the extremities. After treatment of the primary tumor, 40 % to 60% of the patients will develop local or distant recurrent disease. The ultimate determinant of survival in patients with bone and soft tissue sarcomas is the development of distant metastasis. Modern multimodality therapy has improved patient survival; hence follow-up surveillance strategies are becoming increasingly important with significant clinical and fiscal implications. However, the ideal postoperative protocol vis a vis frequency and appropriate screening modalities for these uncommon neoplasms remains ill-defined. Although guidelines have been proposed for follow-up of patients , there is a paucity of data in medical literature on the effectiveness of these recommendations. A prospective randomized controlled trial to evaluate the effectiveness of follow up strategies in picking up disease recurrence and their role in influencing overall survival would go a long way in answering some of these questions.

DETAILED DESCRIPTION:
Follow up studies are performed for a variety of reasons. The detection of a recurrence of the index lesion is the foundation of surveillance. Detection of other medical conditions is a secondary benefit. Psychologically , follow up testing can serve as a source of reassurance. Whether an increased frequency of follow up and the use of various expensive imaging modalities for screening and early detection of recurrence actually results in improving overall survival of patients with extremity bone and soft tissue sarcomas is a question that remains as yet unanswered. Currently followed post operative surveillance regimes are empirical and vary widely from centre to centre. Allocation of limited health funding should be guided by evidence based recommendations rather than empirical beliefs. An ideal surveillance regime should meet the criteria of easy implementation, accuracy and cost effectiveness.

This study attempts to outline guidelines regarding the role of follow up vis a vis frequency and the use of various imaging modalities for early detection of recurrence in improving overall survival of patients with extremity bone and soft tissue sarcomas . In a vast country like India where patients often travel thousands of kilometers in their search for quality medical care the frequency of routine follow up visits is as important as studying the role of expensive screening modalities while drawing up guidelines for cost effective follow up strategies. Though it is well accepted that in bone and soft tissue sarcomas the majority of recurrences either local or distant would occur in the first two years there has been no study to gauge the effectiveness of an intensive three monthly follow up during this initial "risk" period in improving overall survival . We have therefore further attempted to stratify the patients in both arms into Group A and Group B. Compared to Group A patients, Group B patients would have two less follow up visits per year in the initial two years of follow up. This could help to further reduce both the cost and loss of working man hours in these patients.

Correlation between local failure and the development of metastatic disease remains controversial. Though Lewis et al have suggested that there is strong association of local recurrence with the development of subsequent metastasis and tumor mortality, various prospective randomized trials have failed to show that better local control improves survival.

Though an MRI is advantageous in the initial evaluation of STS its utility in the diagnosis of patients with recurrent lesions, including its comparison with physical examination alone has yet to be documented. Distortion of the anatomy and fibrosis because of prior surgery and radiotherapy makes interpretation of post operative images difficult. In a series of 150 patients from the Rosewall Park Cancer Institute almost all the local recurrences were detected on physical examination and 86% of these were deemed resectable .Does an MRI actually help in the accurate early detection of local recurrence and if so does this early detection and subsequent intervention impact on overall survival? Its use has to be assessed critically with regard to cost effectiveness and efficacy.

Patients with extremity bone and soft tissue sarcomas are more likely to have distant metastasis as their initial site of recurrence . Pulmonary metastasis comprises most of these distant failures. The benefit of detection of recurrence depends on the availability of therapeutic interventions that can prolong survival. The occurrence rate of isolated pulmonary metastasis is in the range of 20% to 40% and there is a potential to salvage these patients. Though Huth et al felt that the impact of resection of pulmonary metastasis on improving survival of patients with soft tissue sarcoma was minimal a retrospective study by Geel et al recommended surgical excision of lung metastasis in order to improve survival. CT scanning of the chest is known to be more sensitive than CXR in detecting lung lesions but its specificity in detecting metastatic lesions is lower. The role of CT scanning in the surveillance of metastatic disease is therefore not clear. Whooley et al do not recommend CT scanning of the chest as a surveillance technique because of the high accuracy of CXR in recurrence detection in their series .

There is enough evidence in literature from other solid tumor types i.e. breast cancer, colorectal cancer and melanoma that challenges the usefulness of multiple follow up imaging tests in terms of efficacy , cost effectiveness and survival benefit .Whether the same surmise holds true for extremity soft tissue sarcoma is a matter of debate. Kane states that for soft tissue sarcomas, patient education and follow up visits with thorough history and physical examination will detect the vast majority of recurrent disease . Goel in his article on "Costs of follow-up after potentially curative treatment for extremity soft-tissue sarcoma" states that several guidelines have been proposed for extremity soft-tissue sarcoma patient follow-up. Literature has yet to reflect the consensus these guidelines suggest and he stresses the need for clinical trials to identify an optimal surveillance strategy, one balancing gains in survival, quality of life, costs, and societal willingness to expend resources .

A prospective randomized controlled trial to evaluate the effectiveness of follow up strategies and their role in influencing overall survival could help in outlining a rational, accurate, easily applicable, cost effective surveillance regime.

ELIGIBILITY:
Inclusion Criteria:

1. Patients operated for primary or recurrent extremity bone & soft tissue sarcomas.(both limb salvage and amputations)
2. Non Metastatic at presentation.
3. Patients reliable for follow-up.

Exclusion Criteria:

1. Non-extremity sarcomas.
2. Metastatic at presentation
3. Patients unreliable for follow up.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500 PATIENTS OVERALL. 250 PATIENTS ON INTENSIVE GROUP 250 PATIENTS ON COST EFFECTIVE GROUP
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 10 years
  Patient survival

SECONDARY OUTCOMES:
Disease free survival | 10 years
  Local or distant recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Dr AJAY PURI, ORTHOPAEDIC ONCOLOGIST, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Cipriano CA, Jang E, Tyler W. Sarcoma Surveillance: A Review of Current Evidence and Guidelines. J Am Acad Orthop Surg. 2020 Feb 15;28(4):145-156. doi: 10.5435/JAAOS-D-19-00002. PMID 31651565
- [Background] Chiesa AM, Spinnato P, Miceli M, Facchini G. Radiologic Assessment of Osteosarcoma Lung Metastases: State of the Art and Recent Advances. Cells. 2021 Mar 4;10(3):553. doi: 10.3390/cells10030553. PMID 33806513
- [Background] Heinemann M, Ranft A, Langer T, Jurgens H, Kreyer J, Vieth V, Schafers M, Weckesser M, Simon T, Hassenpflug W, Corbacioglu S, Bielack S, Mayer-Steinacker R, Kuhne T, van den Berg H, Gelderblom H, Bauer S, Stegger L, Dirksen U. Recurrence of Ewing sarcoma: Is detection by imaging follow-up protocol associated with survival advantage? Pediatr Blood Cancer. 2018 Jul;65(7):e27011. doi: 10.1002/pbc.27011. Epub 2018 Feb 26. PMID 29480574